CLINICAL TRIAL: NCT04983563
Title: Assessment of Actigraphy in the Management of Neonatal Opioid Abstinence Syndrome of Hospitalized Newborn in Intensive Care Units
Brief Title: Actigraphy and Neonatal Abstinence Syndrome of Hospitalized Newborn in Intensive Care Units
Acronym: ACTINEO2
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Caen (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: Elodie LECORPS
Record Dates: First submitted 2021-06-10; First posted 2021-07-30 (Actual); Last update posted 2021-07-30 (Actual); Status verified 2021-05

CONDITIONS: Neonatal Abstinence Syndrome
MeSH Terms: conditions — Neonatal Abstinence Syndrome | interventions — Actigraphy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Actigraphy (Experimental)
  Interventions: Device: Actigraphy, eTact

INTERVENTIONS:
Device: Actigraphy, eTact — Actigraphy will be realized twice a day during 30 minutes and Lipsitz scoring system will be realized at the same moment to analyze the correlation between Lipsitz scoring system and actigraphy.

SUMMARY:
The aim of this study is to analyse the correlation between actigraphy and Lipsitz scoring system in neonatal opioid abstinence syndrome of hospitalized newborn in intensive care units

DETAILED DESCRIPTION:
Hospitalized newborn in intensive care units can receive opioids to manage pain or sedation. Neonatal opioid abstinence syndrome can occur when newborn receive opioid treatment for a long time.

Many scoring systems, like Lipsitz scoring system, are used to diagnose and manage neonatal abstinence syndrome but they are subjective. The majority of items in these scores are motor skills items.

Actigraphy allows to measure objectively the newborn motricity. This study will analyse the correlation between actigraphy and Lipsitz scoring system.

ELIGIBILITY:
Inclusion Criteria:

* Newborn > 22 gestation weeks
* Hospitalization in neonatal intensive care unit at CHU de Caen.
* Opioids treatment > 48 hours.

Exclusion Criteria :

* ante or post-natal brain injury diagnosis
* upper arm motor deficit
* palliative care

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2021-03-01 (Actual); Primary Completion 2022-12-31 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Correlation between actigraphy and Lipsitz scoring system | 7 days
  Actigraphy and Lipsitz scoring system are realized at the same time twice a day

CONTACTS AND LOCATIONS:
Overall Officials: Elodie EL LECORPS, Principal Investigator — CHU CAEN
Locations (1):
- Caen University Hospital, Caen, France

IPD SHARING:
Plan to Share IPD: No